CLINICAL TRIAL: NCT04306016
Title: The Effects of a Model-based Sensory Stimulation Intervention on Preventing Delirium Among Intensive Care Unit Patients: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Liang Surui, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019.521
Record Dates: First submitted 2020-03-08; First posted 2020-03-12 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Delirium, Intensive Care Unit, Randomised Controlled Trial
Keywords: Delirium, sensory stimulation, intensive care unit, prevention
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: An assessor-blinded two-arm randomised controlled trial (RCT) will be conducted.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be blinded to the group allocation and will not be involved in data analysis and results reporting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory stimulation (Experimental): Participants allocated to the intervention group will receive a model-based sensory stimulation intervention, which is aimed at providing visual and auditory stimulation to ICU patients with additional support from family caregivers.
  Interventions: Other: Sensory stimulation
- Usual care (No Intervention): Participants in the control group will receive usual care routine that they are receiving or planning to receive. The registered ICU nurses will provide the same nursing care as previously, including but not limiting to the use of sedation, analgesia, spontaneous breathing trial, indwelling catheter, feeding, and bowel care.

INTERVENTIONS:
Other: Sensory stimulation — Sensory stimulation can be formed in different aspects, and the most important ones are visual stimulation and auditory stimulation. Visual stimulation interventions involved providing a calendar, clock or familiar objects such as photographs of family caregivers; while auditory stimulation included calling the name of patients, helping to orientate the time and location, introducing hospital information, the ICU surrounding and treatment, and communicating with patients, who could not talk due to artificial airway, through a blackboard and use of gestures.
  Arms: Sensory stimulation

SUMMARY:
Delirium is highly associated with adverse clinical outcomes of intensive care unit (ICU) patients, including increased cognitive impairment, duration of intubation, ICU length of stay, mortality, physical dependence, and health care costs. This randomised controlled study will firstly develop a family-supported sensory stimulation package based on the literature review as well as the findings of the cross-sectional survey and the in-depth interview. The intervention effects than will be evaluated using outcomes including delirium incidence, delirium duration, delirium severity, ICU patients' consciousness and cognitive function as well as family members' satisfaction and anxiety. This study is expected to provide evidence of the effectiveness of family-supported sensory stimulation on preventing delirium among ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* the first time admitted to ICU
* a Richmond Agitation-Sedation Scale (RASS) score ≥-3

Exclusion Criteria:

* diagnosed with stroke, dementia, delirium or acute psychiatric illness at admission
* diagnosed with end-stage of cancer
* severe hearing impairment and cannot be corrected by hearing aids
* admitted to ICU with radiative material.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Delirium incidence | Through study completion, an average of seven days
  Delirium incidence means the number of patients who are delirious.
First occurrence of delirium | Through study completion, an average of seven days
  First occurrence of delirium was defined as the first time that patients was delirium positive through CAM-ICU. The time to have the first occurrence of delirium was calculated from patients' admission to ICU to the first positive result of delirium assessment.
Delirium duration | Through study completion, an average of seven days
  The delirium duration will be calculated when the patient is first considered to have delirium to the last time that patient is not supposed to have delirium based on CAM-ICU.
Delirium severity | Through study completion, an average of seven days
  CAM-ICU-7 scores are further categorised as 0-2: no delirium, 3-5: mild to moderate delirium, and 6-7: severe delirium.

SECONDARY OUTCOMES:
Post-traumatic stress disorder (PTSD) | Through study completion, an average of seven days
  The 17-item PTSD Checklist (PCL) correspond to the DSM-III-R symptoms of PTSD (post-traumatic stress disorder), which is a self-reporting scale for assessing PTSD (Frank et al., 1993; Mollica et al., 1992). Patients were asked for their agreement to describe each item, from one (not at all) to five (extremely). PTSD-symptoms could be divided into re-experiencing (flashback, nightmare, emotional cue reactivity, and physical cue reactivity), avoidance and emotional numbing (avoidance of thoughts and reminders, amnesia, loss of interest, detachment, restricted affect, and foreshortened future) and hyperarousal (irritability/anger, sleep disturbance, difficulty concentrating, hypervigilance, exaggerated startle response). The total score was summed and ranged from 17 to 85
Depressive symptoms | Through study completion, an average of seven days
  The 9-item Chinese version of Patient Health Questionnaire-9 (PHQ-9) will be used to measure patients' psychological well-being.Patients will be asked for their agreement to the description of each item, from zero (not at all) to three (nearly every day). All item scores are summed (total score = 27). A higher score indicates greater severity of the depressive symptoms.
Family satisfaction | Through study completion, an average of seven days
  Family satisfaction will be measured using the Critical Care Family Satisfaction Survey (CCFSS).CCFSS has 27 items and five dimensions: medical condition guarantee, access to information, acceptance, support, and comfort. Family caregivers will be asked for their agreement to the description of each item, from one (very unsatisfactory) to five (very satisfactory). All item scores are summed (total score = 135). A higher score indicates a greater level of satisfaction.
Level of anxiety | Through study completion, an average of seven days
  The level of anxiety of family caregivers will be measured by the Self-Rating Anxiety Scale (SAS). SAS has 20 items, with each item ranging from one (not at all) to four (very much so). The scale will use both positive and negative scoring, with a total score of 50-59 indicating mild anxiety, 60-69 indicating moderate anxiety, and ≥70 indicating severe anxiety.
ICU memory | Through study completion, an average of seven days
  The ICU-Memory Tool (ICU-M) was used to measure ICU patients' ICU experience (Jones et al., 2000). The tool includes 14 questions (five open-ended questions and nine closed-ended questions), mainly including three parts: memories before admission to ICU; memories during ICU stay and memories after transferring out of ICU. Memories during ICU stay has three subscales: factual memories (lights, alarms, voices, families, faces, breathing tube, suctioning, darkness, clock, tube in your mouth, and ward wounds), memories of feelings (being uncomfortable, confused, down, anxious/ frightened, panic, and pain), and memories of delusions (feeling that people were trying to hurt you, hallucinations, nightmares, dreams). We summed the number of memories in each of the three subscales. The Chinese version of ICU-M has a Cronbach α coefficient of 0.823 and a scale-level content validity index of 0.946, which confirms its good reliability and validity
Depressive symptoms | At one month upon patients' admission to ICU
  The 9-item Chinese version of Patient Health Questionnaire-9 (PHQ-9) will be used to measure patients' psychological well-being.Patients will be asked for their agreement to the description of each item, from zero (not at all) to three (nearly every day). All item scores are summed (total score = 27). A higher score indicates greater severity of the depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China